CLINICAL TRIAL: NCT04557839
Title: Effects of Balance Training on Vestibular Function and Proprioception Feedback in Stroke Patient
Brief Title: Balance Training on Vestibular Function and Proprioception Feedback in Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/20/2050 Asia bashir
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Stroke, Ischemic
Keywords: Balance training; Stroke; Proprioceptive feedback; Vestibular function
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy balance exercise (Active Comparator): Traditional physical therapy including balance exercise on mate and swiss ball.
  Interventions: Other: Traditional physical therapy balance exercise
- proprioception based balance training (Experimental): proprioception based balance training with eye open and close on soft , firm and foam surface.
  Interventions: Other: proprioception based balance training

INTERVENTIONS:
Other: Traditional physical therapy balance exercise — first phase : stepping forward, backward, and sideways on the exercise step stepping over blocks of various heights standing up from a chair, walking four steps forward,)A performing a range of motion and balance exercises (forward and backward rolling of the arms; bending the trunk forward and side to side);on a swiss ball. performed In a normal condition In first 20 m of each session 2nd phase Performing double-legged stance tandem walking forward and backward
  • Dosage of exercise was twice a week for 6 week each session comprise of 60 mints. Each set consisted of 4 periods of 11 exercises and rest of 40 sec .many exercise over time will turn into circuit training
  Arms: Traditional physical therapy balance exercise
Other: proprioception based balance training — first phase : stepping forward, backward, and sideways on the exercise step stepping over blocks of various heights standing up from a chair, walking four steps forward,)A performing a range of motion and balance exercises (forward and backward rolling of the arms; bending the trunk forward and side to side);on a swiss ball. performed In a normal condition In first 20 m of each session 2nd phase Performing double-legged stance tandem walking forward and backward all exercise done under following condition.
  * eyes open firm surfaces
  * Eyes open soft surfaces
  * Eyes closed firm surfaces
  * Eyes closed soft surfaces (the soft surfaces will be a foam mate with 2.5 cm thick )
  * These exercise will perform with turning the head side to side ad up and down
  * Dosage of exercise was twice a week for 6 week each session comprise of 60 mints. Each set consisted of 4 periods of 11 exercises and rest of 40 sec .many exercise over time will turn into circuit training
  Arms: proprioception based balance training

SUMMARY:
The aim of this study was to find out the role of balance training on vestibular function and proprioception feedback in stroke patients. It was a randomized control trial and was conducted in civil hospital Gujranwala. Current study was completed within the time duration of 6 month. Sample size of twenty four patient consists of both male and female aged between 50 years to 75 years. Each group contain 12 patient .Group A was experimental group which received balance exercise in two phases and group B (n=12) was control group received conventional therapy. Each of exercise program begun with 10 mints warm up consisting of walking ad light stretching of hip flexor. The balance training group received the balance training exercise twice a week for 6 week each session comprise of 60 minutes. Each set consisted of 4 periods of 11 exercises and rest of 40 seconds. Many exercises over time was turned into circuit training. Data was analyzed by using SPSS version 23.

DETAILED DESCRIPTION:
Stroke is a global health-care problem that is common, serious, and disabling in most countries, the 2nd or 3rd most common cause of death and one of the main causes of acquired adult disability. Patients with stroke have number of impairments but usually present with difficulty maintaining balance. Balance is described as the ability to maintain equilibrium in a gravitational field by keeping or returning the center of body mass over its base of support. Body balance is the result of a harmonious interaction between the afferents from sensory systems (vestibular, proprioceptive and visual). The somatosensory system organizes proprioceptive information, while the visual system provides information about the position of the body in relation to the external environment. When the functions of the sensory triad are disrupted, unpleasant sensations occur, e.g. dizziness, nausea, feeling of imbalance and, sometimes, nystagmus, Balance is a complex process in which the maintenance of a position is regulated by postural adjustments to voluntary activity and in response to external perturbation. Impairments of postural control result in increased rates of unintentional falls. In fact, falls are the leading cause of injuries and subsequent deaths among people 65 years and older, and generate a fundamental financial burden to the healthcare system.Stroke survivors present with deficits in different systems, including sensory, musculoskeletal, perceptual, and cognitive, which decrease postural stability. The lack of postural stability can lead to falls during hospitalization, both in the acute care and rehabilitation stages, and after discharge. Because of the importance of postural instability in this population, a systematic evaluation of balance is needed to identify specific problems.The measures most commonly used with stroke patients are different parameters extracted from the center of pressure (COP) and weight distribution of the vertical reaction force. After a stroke, patients have demonstrated a significant increase in sway and weight-bearing asymmetry. The relearning of postural control through external visual and auditory biofeedback is believed to be an effective therapy for improving balance control. In a Cochrane review, the results of seven randomized clinical trials and indicated that providing feedback from a force platform resulted in improved stance symmetry after stroke but did not improve balance during active functional activities, nor did it improve overall independence. A study conducted on elderly population was concluded that Balance training reduced elderly subjects' overactive proprioceptive feedback and enhanced vestibular orientation Previous studies only assess the effect of balance training on elderly population or stroke population. But the role of these trainings on vestibular and proprioception function were not assessed among stoke population while in the current study we aimed to assess the effect of balance training of simple physical therapy exercises on sensory channel (vestibular function, proprioception feedback mainly). In 2011 on Stroke rehabilitation was concluded by Ongoing trials of repetitive task training, early mobilization, treadmill training, physical fitness training, and speech and language training for aphasia and dysarthria are high-quality, multicenter, multidisciplinary studies of complex interventions, which meet many of the above recommendations.

In 2004 a comparative study to compare clinical and biomechanical measures of balance in elderly stroke patients with those of healthy elderly people. This study concluded as postural stability in quiet stance, as measured by COP-COM amplitude, was related to functional measures of balance as well as physiologic factors relating to balance, such as visual conditions, lower-extremity peripheral sensibility, motor recovery, and simple reaction time Another study on dynamic balance ability through stair gait training where in proprioceptive neuromuscular facilitation (PNF) was applied and for the four weeks of the experiment, each group received training three times per week, for 30 min each time. Berg Balance Scale (BBS) values were measured and a time up and go (TUG) test and a functional reach test (FRT) were performed for a comparison before and after the experiment which is concluded that gait training group to which PNF was applied saw improvements in their balance ability, and a good result is expected when neurological disease patients receive stair gait training applying PNF.(10) A systematic review evaluated recent evidence related to the effect of balance training on balance performance among individuals post stroke across the continuum of recovery. On the basis of this evidence, we also provide recommendations for exercise prescription in such programs. Review evaluated recent evidence related to the effect of balance training on balance performance among individuals post stroke across the continuum of recovery. On the basis of this evidence, we also provide recommendations for exercise prescription in such programs.

In 2o18 on to investigate the effect of customized vestibular rehabilitation training on gait stability of patients with sub-acute stroke. An instrumented 10- Meter Walk Test together with traditional clinical scales were used to assess VR effects. Which is concluded by VR could be included into a rehabilitation program for patients with stroke for improving their gait and dynamic balance acting on their vestibular system as facilitator of recovery.

Another study in 2014 virtual reality (VR) proprioception rehabilitation system was developed for stroke patients to use proprioception feedback in upper limb rehabilitation by blocking visual feedback. To evaluate its therapeutic effect, 10 stroke patients (onset > 3 month) trained proprioception feedback rehabilitation for one week and visual feedback rehabilitation for another week in random order. Proprioception functions were checked before, a week after, and at the end of training.it was concluded that effectiveness and possible use of the VR to recover the proprioception of stroke patients In 2020 A pilot study to find out the effects of COP (center of pressure) movement tracking training conducted using the Biodex Balance System SD in static and dynamic modes on balance ability in stroke patients. The result of study concluded that COP movement tracking training in dynamic mode was found to be a more effective intervention for improving the static balancing abilities of stroke patients than training in static mode.

In 2000 A comparative study was done by walker et al to compared the relative effectiveness of visual feedback training of center-of-gravity (COG) positioning with conventional physical therapy following acute stroke result show that Visual feedback or conventional balance training in addition to regular therapy affords no added benefit when offered in the early stages of rehabilitation following stroke

ELIGIBILITY:
Inclusion Criteria:

* Participants with impaired balance ,vestibular function and proprioception due to stroke
* Victim of a stroke that resulted in hemiparesis,
* Be at least 6 months
* Be fully discharged from all rehabilitation program

Exclusion Criteria:

* Those with recurrent strokes
* Bilateral hemispheric cerebellar or brain stem lesions
* Severe spasticity or cognitive deficit
* Orthopedic or peripheral neuropathy
* Significant visual field or hemi neglect problems were excluded.
* They were medically unstable as determined by examination, history, or medical records.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Fukuda stepping test | 6 week
  Changes from the baseline, It is neurological test to test vestibular function. Patient was asked to take 50 steps withy eyes closed in circle. After 50nsteps angle and distance measured from the initial to terminal position.
Berg Balance Scale | 6 week
  Changes from the baseline, The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. A score of 56 indicates functional balance.A score of < 45 indicates individuals may be at greater risk of falling

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Civil hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pimentel BN, Filha VAVDS. Evaluation of vestibular and oculomotor functions in individuals with dizziness after stroke. Arq Neuropsiquiatr. 2019 Jan;77(1):25-32. doi: 10.1590/0004-282X20180154. PMID 30758439
- [Background] Wiesmeier IK, Dalin D, Wehrle A, Granacher U, Muehlbauer T, Dietterle J, Weiller C, Gollhofer A, Maurer C. Balance Training Enhances Vestibular Function and Reduces Overactive Proprioceptive Feedback in Elderly. Front Aging Neurosci. 2017 Aug 11;9:273. doi: 10.3389/fnagi.2017.00273. eCollection 2017. PMID 28848430
- [Background] Corriveau H, Hebert R, Raiche M, Prince F. Evaluation of postural stability in the elderly with stroke. Arch Phys Med Rehabil. 2004 Jul;85(7):1095-101. doi: 10.1016/j.apmr.2003.09.023. PMID 15241756
- [Background] Barclay-Goddard R, Stevenson T, Poluha W, Moffatt ME, Taback SP. Force platform feedback for standing balance training after stroke. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD004129. doi: 10.1002/14651858.CD004129.pub2. PMID 15495079
- [Background] Yavuzer G, Eser F, Karakus D, Karaoglan B, Stam HJ. The effects of balance training on gait late after stroke: a randomized controlled trial. Clin Rehabil. 2006 Nov;20(11):960-9. doi: 10.1177/0269215506070315. PMID 17065539
- [Background] Seo K, Park SH, Park K. The effects of stair gait training using proprioceptive neuromuscular facilitation on stroke patients' dynamic balance ability. J Phys Ther Sci. 2015 May;27(5):1459-62. doi: 10.1589/jpts.27.1459. Epub 2015 May 26. PMID 26157240
- [Background] Lubetzky-Vilnai A, Kartin D. The effect of balance training on balance performance in individuals poststroke: a systematic review. J Neurol Phys Ther. 2010 Sep;34(3):127-37. doi: 10.1097/NPT.0b013e3181ef764d. PMID 20716987
- [Background] Tramontano M, Bergamini E, Iosa M, Belluscio V, Vannozzi G, Morone G. Vestibular rehabilitation training in patients with subacute stroke: A preliminary randomized controlled trial. NeuroRehabilitation. 2018;43(2):247-254. doi: 10.3233/NRE-182427. PMID 30040765
- [Background] Cho S, Ku J, Cho YK, Kim IY, Kang YJ, Jang DP, Kim SI. Development of virtual reality proprioceptive rehabilitation system for stroke patients. Comput Methods Programs Biomed. 2014;113(1):258-65. doi: 10.1016/j.cmpb.2013.09.006. Epub 2013 Sep 19. PMID 24183070
- [Background] Cha JH, Kim NH, Cha YJ. Effect of proprioceptive stimulation induced by footplate during center of pressure movement tracking training on the balance abilities of patients with chronic hemiplegic stroke: a randomized, controlled, pilot study. Top Stroke Rehabil. 2020 Jan;27(1):38-43. doi: 10.1080/10749357.2019.1661699. Epub 2019 Sep 4. PMID 31480897
- [Background] Smania N, Picelli A, Gandolfi M, Fiaschi A, Tinazzi M. Rehabilitation of sensorimotor integration deficits in balance impairment of patients with stroke hemiparesis: a before/after pilot study. Neurol Sci. 2008 Oct;29(5):313-9. doi: 10.1007/s10072-008-0988-0. Epub 2008 Oct 21. PMID 18941933
- [Background] Mao Y, Chen P, Li L, Huang D. Virtual reality training improves balance function. Neural Regen Res. 2014 Sep 1;9(17):1628-34. doi: 10.4103/1673-5374.141795. PMID 25368651
- [Background] Walker C, Brouwer BJ, Culham EG. Use of visual feedback in retraining balance following acute stroke. Phys Ther. 2000 Sep;80(9):886-95. PMID 10960936
- [Background] Chen IC, Cheng PT, Chen CL, Chen SC, Chung CY, Yeh TH. Effects of balance training on hemiplegic stroke patients. Chang Gung Med J. 2002 Sep;25(9):583-90. PMID 12479619
- [Background] Donath L, Roth R, Zahner L, Faude O. Slackline Training (Balancing Over Narrow Nylon Ribbons) and Balance Performance: A Meta-Analytical Review. Sports Med. 2017 Jun;47(6):1075-1086. doi: 10.1007/s40279-016-0631-9. PMID 27704483